CLINICAL TRIAL: NCT05021718
Title: Effectiveness of Strengthening Exercise Plus Activities of Daily Living Instructions in Reducing Pain in Patients With Lumbar Disc Herniation
Brief Title: Strengthening Exercise and Activities of Daily Living Instructions for Patients With Lumbar Disc Herniation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chittagong Medical College (Other)
Responsible Party: Principal Investigator, MD Imam Shahriar, FCPS student, Chittagong Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LDH exercise
Record Dates: First submitted 2021-08-22; First posted 2021-08-25 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Lumbar Disc Herniation
Keywords: Low back pain; Disc herniation; Strengthening exercise; ADL instructions
MeSH Terms: conditions — Intervertebral Disc Displacement; Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (IG) (Experimental): A total of 35 patients in IG received different back and hip strengthening exercises five times a week for six weeks. They were also instructed to follow the ADLIs to perform different tasks at home and in workplaces during the intervention and at least 3 months after the intervention.
  Interventions: Other: Strengthening exercises; Behavioral: Activities to daily living instructions
- Control group (CG) (Active Comparator): The remaining 35 patients were allocated to CG. The patients in CG were treated with Naproxen (500 mg) and Baclofen (10 mg) tablet twice a day for three weeks, followed by hot moist compression for the next three weeks. Moreover, they were instructed to follow the ADLIs to perform different tasks at home and in workplaces during the intervention and at least 3 months after the intervention.
  Interventions: Drug: Pharmacological therapy; Other: Hot compression; Behavioral: Activities to daily living instructions

INTERVENTIONS:
Other: Strengthening exercises — Back and hip strengthening exercises. The intensity of exercises was based on the exercise tolerance and pain thresholds of the individual subjects.
  Arms: Intervention group (IG)
Drug: Pharmacological therapy — Naproxen (500 mg) and Baclofen (10 mg) tablet twice a day for three weeks
  Arms: Control group (CG)
Other: Hot compression — Hot moist compression from week 4 to week 6.
  Arms: Control group (CG)
Behavioral: Activities to daily living instructions — * Avoid forward bending.
  * Avoid heavy weightlifting.
  * Avoid prolong standing.
  * Avoid prolong sitting.
  * Use a plain firm bed.
  * Lie down in a supine position.

SUMMARY:
Lumbar disc herniation (LDH) is one of the most common causes of mechanical low back pain (LBP) associated with radiating leg pain. Conservative treatment, including exercise, analgesic, and physical therapy, is regarded as the first-line treatment of LDH.

This randomized clinical trial was conducted to evaluate the effectiveness of back and hip strengthening exercises combined with activities of daily living instructions (ADLIs) to reduce pain intensity in patients with LDH.

DETAILED DESCRIPTION:
A total of 70 patients with LDH were randomly allocated to either the intervention group (IG) or the control group (CG). Patients in IG received different back and hip strengthening exercises five days a week for six weeks. The patients in CG were treated with Naproxen (500 mg) and Baclofen (10 mg) tablet twice a day for three weeks, followed by hot moist compression for the next three weeks. In addition, the patients in both groups were instructed to follow the ADLIs during the intervention and at least 3 months after the intervention.

The straight leg raising (SLR) test and the Visual Analogue Scale (VAS) score were used to evaluate the patients' pain intensity. Outcomes were measured at baseline, at three weeks, and six weeks of the intervention. Patients were followed up after 3 months of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 59 years.
* Clinically diagnosed LDH that was confirmed by MRI.
* Duration of the pain: ≥ 3 months

Exclusion Criteria:

* Painful spinal deformity
* Cauda equina syndrome
* Progressive neurological signs and/or muscle-wasting
* History of spinal surgery, spine fracture, scoliosis, tuberculosis, and tumours.
* Treated with epidural injections.
* Pregnancy

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Changes in perceived pain intensity | Outcomes were evaluated at baseline, at three weeks, and six weeks of the intervention. Patients were followed up after 3 months of the intervention.
  Visual analog scale (VAS) score: Patients were asked to rate their perceived pain on a 0-to-10-point scale, where 0 indicated no pain at all and 10 indicated the most severe imaginable pain.

SECONDARY OUTCOMES:
Changes in the range of hip flexion during straight leg raising test | Outcomes were evaluated at baseline, at three weeks, and six weeks of the intervention. Patients were followed up after 3 months of the intervention.
  The range of hip flexion during affected and unaffected straight leg raising without pain was measured by hand-held goniometry.

CONTACTS AND LOCATIONS:
Locations (1):
- Chittagong Medical College Hospital, Chittagong, Bangladesh

IPD SHARING:
Plan to Share IPD: No